CLINICAL TRIAL: NCT00600756
Title: A One-Year Randomized, Prospective, Parallel, Open Comparison of Subjective Well-being in Schizophrenic Out-patients Treated With Quetiapine XR (SEROQUEL XR™) or Oral Risperidone at Flexible Dose in a Naturalistic Setting
Brief Title: Comparison of the Subjective Well-being and Tolerability of Quetiapine XR to Risperidone
Acronym: RECOVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00039
Record Dates: First submitted 2008-01-09; First posted 2008-01-25 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Schizophrenic Disorders
Keywords: schizophrenia; SWNK
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

ARMS (2):
- Quetiapine XR (Experimental)
  Interventions: Drug: Quetiapine XR
- Risperidone (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Quetiapine XR — Oral, once daily, tablets of 400 mg to 800 mg
  Other Names: Seroquel XR
  Arms: Quetiapine XR
Drug: Risperidone — Oral, once daily, tablets of 2 mg to 6 mg
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
The trial is designed to assess the long term subjective well-being in schizophrenic outpatients treated with quetiapine XR (extended release) or oral risperidone at flexible dose in a naturalistic setting over a period of one year. Secondary outcome measures have been selected for helping in the differentiation of the compared atypical antipsychotics. The primary objective of this study is to demonstrate the non-inferiority of quetiapine XR to risperidone assessed at month 6 in terms of responder rate using the self-report instrument SWN-K

ELIGIBILITY:
Inclusion Criteria:

* Treated for symptomatic schizophrenia (DSM-IV-TR codes: 295.10, 295.20, 295.30,295.60, 295.90) or schizoaffective disorder (DSM-IV-TR code:295.70) or schizophreniform disorder (DSM-IV-TR code: 295.40). Patients with co-morbid depressive symptoms may be enrolled
* Patient with first episode of the above mentioned disease (item 3) or patient requiring a medication change for clinical reasons (effectiveness, tolerability, compliance, patient preference), i.e. switch from typical to atypical neuroleptics, switch from other atypical neuroleptics, excluding patients treated with risperidone or quetiapine at the time of enrolment.

Exclusion Criteria:

* Patients with a baseline SWN-K total score of >75
* Patients with previous treatment with risperidone or quetiapine may be enrolled if change of treatment has not been dictated by major lack of tolerability and efficacy and if date of last dose has been at least 3 months prior to enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brecher, MSD, Study Director — AstraZeneca; Prof Naber, MD, Principal Investigator — Klinikum Eppendorf
Locations (116):
- Belgium (7):
  - Research Site, Assebroek, Belgium
  - Research Site, Hasselt, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Montignies-sur-Sambre, Belgium
  - Research Site, Roeselare, Belgium
  - Research Site, Sint-Denijs-Westrem
  - Research Site, Tournai
- Brazil (13):
  - Research Site, Fortaleza, Ceará
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Aparecida de Goiânia, Goiás
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Itapira, São Paulo
  - Research Site, Ribeirão Preto, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Sorocaba, São Paulo
  - Research Site, Botucatu
- Bulgaria (7):
  - Research Site, Cerova Koria Village, Veliko Tarnovo
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Costa Rica (3):
  - Research Site, Barrio Los Yoses, Provincia de San José
  - Research Site, Curridabat, Provincia de San José
  - Research Site, Guadalupe, Provincia de San José
- Finland (9):
  - Research Site, Helsinki
  - Research Site, Kitee
  - Research Site, Kuopio
  - Research Site, Lapua
  - Research Site, Pori
  - Research Site, Raahe
  - Research Site, Rovaniemi
  - Research Site, Tampere
  - Research Site, Turku
- Germany (20):
  - Research Site, Bad Saarow
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bochum
  - Research Site, Butzbach
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Duisburg
  - Research Site, Gelsenkirchen
  - Research Site, Grevenbroich
  - Research Site, Hamburg
  - Research Site, Hattingen
  - Research Site, Hildesheim
  - Research Site, Königsbrück
  - Research Site, Mittweida
  - Research Site, München
  - Research Site, Oranienburg
  - Research Site, Siegen
  - Research Site, Stralsund
  - Research Site, Wismar
- Italy (16):
  - Research Site, Andria, BA
  - Research Site, Feltre, BL
  - Research Site, Maddaloni, CE
  - Research Site, Sora, FR
  - Research Site, Genova, GE
  - Research Site, Milan, MI
  - Research Site, Perugia, PG
  - Research Site, Fidenza, PR
  - Research Site, Parma, PR
  - Research Site, Palmi, RC
  - Research Site, Rimini, RN
  - Research Site, Salerno, SA
  - Research Site, Sassari, SS
  - Research Site, Chioggia, VE
  - Research Site, Ancona
  - Research Site, Pompei
- Mexico (7):
  - Research Site, México, D.f.
  - Research Site, México, D.F
  - Research Site, Monterrey, Nuevo Leon, Mexico
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Guadalajara Jalisco
  - Research Site, México
  - Research Site, Yucatán
- Portugal (6):
  - Research Site, Abraveses
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Santarém
- Romania (5):
  - Research Site, Piteşti, Argeş
  - Research Site, Galati, Galați County
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Sibiu
- Russia (4):
  - Research Site, Moscow, Russia
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (12):
  - Research Site, Jaén, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Zamudio (vizcaya), Basque Country
  - Research Site, Salamanca, Castille and León
  - Research Site, Zamora, Castille and León
  - Research Site, Mataro (barcelona), Catalonia
  - Research Site, Vigo, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Langreo, Principality of Asturias
  - Research Site, Elche (alicante), Valencia
  - Research Site, Sant Joan d'Alacant, Valencia
- Switzerland (2):
  - Research Site, Prilly, Canton of Vaud
  - Research Site, Wil
- Turkey (Türkiye) (5):
  - Research Site, Istanbul, Turkey
  - Research Site, Manisa, Turkey
  - Research Site, Ankara
  - Research Site, Elâzığ
  - Research Site, Izmir

REFERENCES:
- [Derived] Naber D, Peuskens J, Schwarzmann N, Goltz M, Kruger H, Lambert M, Haro JM. Subjective well-being in schizophrenia: a randomised controlled open-label 12-month non-inferiority study comparing quetiapine XR with risperidone (RECOVER). Eur Neuropsychopharmacol. 2013 Oct;23(10):1257-69. doi: 10.1016/j.euroneuro.2013.07.006. Epub 2013 Jul 29. PMID 23953270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a 1-year, randomized, prospective, parallel, open-label study. The study was conducted in 114 study centers in 13 countries.
  OR International multi-center study, 180 sites recruited between January 2008 and October 2009.
Pre-assignment Details: Screening for eligibility. Patients with a SWN-K total score ≤ 75 were entered into the study.
  All patients with "no intake of IP and missing SWN-K total score at baseline or following baseline were included in the study "Overall Number of Participants" but these patients are excluded from the ITT Analysis set!
Groups:
- Quetiapine XR: Experimental - oral, once daily, tablets of 400 mg to 800 mg
- Risperidone: Active Comparator - oral, once daily, tablets of 2 mg to 6 mg
Period: Analysis After 6 Months
Arm/Group | Quetiapine XR | Risperidone
Started | 395 | 403
Completed | 264 (Completers are all patients who completed the study up to Visit 5 (including premature withdraw)) | 283 (Completers are all patients who completed the study up to Visit 5 (including premature withdraw))
Not Completed | 131 | 120
Not completed — Adverse Event | 43 | 33
Not completed — Withdrawal by Subject | 38 | 30
Not completed — Incorrect Enrollment | 12 | 21
Not completed — worsening symptom, lack of efficacy | 11 | 14
Not completed — Severe non-compliance to protocol | 11 | 11
Not completed — Lost to Follow-up | 10 | 8
Not completed — Study-specific discontinuation criteria | 6 | 3
Period: Overall Study Analysis After 12 Months
Arm/Group | Quetiapine XR | Risperidone
Started | 395 | 403
Randomized Analysis | 395 | 403
Safety Analysis | 391 | 402
ITT Analysis | 379 | 392
Completed | 212 (Completed study to Visit 7 (includes premature withdrawals with final visit in the Visit 7 window)) | 227 (Completed study to Visit 7 (includes premature withdrawals with final visit in the Visit 7 window))
Not Completed | 183 | 176
Not completed — Adverse Event | 53 | 44
Not completed — Withdrawal by Subject | 51 | 41
Not completed — Incorrect enrollment | 21 | 29
Not completed — worsening symptom, lack of efficacy | 17 | 20
Not completed — Severe non-compliance to protocol | 16 | 20
Not completed — Lost to Follow-up | 16 | 13
Not completed — Study-specific discontinuation criteria | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Risperidone | Total
Number analyzed (Participants) | 395 | 403 | 798
Age Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (11.7) | 40.0 (11.66) | 39.7 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 171 | 333
  Male | 233 | 232 | 465

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate at Month 6 in the Per Protocol Population Using the Subjective Well-being Under Neuroleptics Scale, Short Version (SWN-K) Total Score
Description: The SWN-K is comprised of 20 questions, rated on a 6-point scale from 1 (not at all) to 6 (very much). Scores range from 20 to 120, with higher scores implying higher subjective well-being. A responder is defined as a subject with an increase of 10 points or 20% from baseline in SWN-K total score (non-inferiority limit of -9.7% in responder rate)
Time Frame: 6 months
Population: For Per Protocol at Month 6 analysis, the difference from Randomized analysis (395) was no study drug (4); SWN-K score missing (12), and did not meet inclusion criteria (169) for Quetiapine XR. For Risperidone, the difference from Randomized analysis (403) was no study drug (1); SWN-K score missing (10), and did not meet inclusion criteria (160).
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 210 | 232
Participants | 136 | 158

2. Secondary Outcome: Change From Baseline in Mean Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Total Score at Month 12 in the Per Protocol Population
Description: The SWN-K is comprised of 20 questions, each of which is rated using a 6-point scale ranging from 1 (not at all) to 6 (very much). Possible scores range from 20 to 120, with higher scores implying higher subjective well-being.
Time Frame: Baseline and Month 12
Population: For Per Protocol at Month 12 analysis, the difference from Randomized analysis (395) was no study drug (4); SWN-K score missing (12), and did not meet inclusion criteria (206) for Quetiapine XR. For Risperidone, the difference from Randomized analysis (403) was no study drug (1); SWN-K score missing (10), and did not meet inclusion criteria (201).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 173 | 191
Scores on a scale | 23.2 (1.55) | 21.1 (1.49)

3. Secondary Outcome: Change From Baseline in Mean Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Total Score at Month 12 in the Intent-to-Treat (ITT) Population
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Scores on a scale | 22.7 (1.34) | 19.4 (1.0)

4. Secondary Outcome: Change From Baseline in the Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Subscale Score: Physical Functioning at Month 12 in the ITT Population.
Description: The SWN-K total score is the sum of 5 subscores (4 questions each): physical functioning, social integration, mental functioning, self-control, and emotional regulation. The subscores are rated using a 6-point scale (the higher the grade, the better the response). Possible subscores range from 4 to 24.
Time Frame: Baseline and 12 months
Population: The ITT analysis set at Month 12 is presented. For Quetiapine XR, there were 168 missing CGI-SCH assessments, resulting in 211 evaluable subjects at Month 12. For Risperidone, there were 165 missing CGI-SCH assessments, resulting in 227 evaluable subjects at Month 12.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Scores on a scale | 4.9 (0.32) | 4.0 (0.31)

5. Secondary Outcome: Change From Baseline in the Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Subscale Score: Social Integration at Month 12 in the ITT Population.
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Scores on a scale | 4.6 (0.32) | 4.0 (0.31)

6. Secondary Outcome: Change From Baseline in the Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Subscale Score: Mental Functioning at Month 12 in the ITT Population.
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Scores on a scale | 4.9 (0.31) | 3.9 (0.30)

7. Secondary Outcome: Change From Baseline in the Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Subscale Score: Self-control at Month 12 in the ITT Population.
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Scores on a scale | 4.1 (0.29) | 3.8 (0.29)

8. Secondary Outcome: Change From Baseline in the Subjective Well-Being Under Neuroleptic Treatment Scale (SWN-K) Subscale Score: Emotional Regulation at Month 12 in the ITT Population.
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Scores on a scale | 4.5 (0.32) | 3.9 (0.31)

9. Secondary Outcome: The Remission Rate in Both the Quetiapine XR Group and the Risperidone Group at Month 12 in the ITT Population
Description: Remission was defined as a SWN-K total score greater than or equal to 80. The reported population is participants who showed remission over, time from baseline to Month 12
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 210 | 227
Participants | 139 | 128

10. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone at Month 12 in the ITT Population on Core Schizophrenic and Depressive Symptoms by Evaluating the Change From Baseline in CGI-SCH Overall Severity Score (Improved).
Description: For the CGI-SCH overall severity of illness, the score ranged from 1 (normal, not ill) to 7 (among the most severely ill). CGI-SCH score was divided into 3 classes: worsening (change score>0), stable (change score=0) and improved (change score<0). Change from baseline in CGI-SCH overall severity of illness in number of participants with CGI-SCH overall severity score improvement.
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 211 | 227
Participants | 176 (1.46) | 178

11. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone at Month 12 in the ITT Population on Core Schizophrenic and Depressive Symptoms by Evaluating the Change From Baseline in CGI-SCH Overall Severity Score
Description: For the CGI-SCH (Clinical Global Impression-Schizophrenia severity of illness scale) overall severity of illness, the score ranged from 1 (normal, not ill) to 7 (among the most severely ill). Change from baseline in CGI-SCH score was divided into 3 classes: worsening (change score>0), stable (change score=0) and improved (change score<0).
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 211 | 227
Scores on a scale | 3.8 (0.63) | 3.9 (0.67)

12. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone at Month 12 in the ITT Population on Core Schizophrenic and Depressive Symptoms by Evaluating the Change From Baseline in the Calgary Depression Scale for Schizophrenia (CDSS) Total Score
Description: The CDSS total score is the sum of 9 questions and ranges from 0 to 27. The higher the score, the more severe are the symptoms.
Time Frame: 12 months
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 351 | 362
Scores on a scale | -4.7 (0.26) | -3.7 (0.25)

13. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone by Evaluating the Relapse Rate at Month 12 in the ITT Population
Description: Relapse is defined as at least one increase of greater than or equal to 2 points on the CGI-SCH overall severity score during the treatment period or at least one hospitalization due to psychiatric disorders during the treatment period.
Time Frame: 12 months
Population: The Reported population is participants who showed relapse over time, from baseline to Month 12.
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Participants | 43 | 31

14. Secondary Outcome: Evaluation of Effect of Quetiapine XR Versus Risperidone on the Health-related Quality of Life of Patients With Schizophrenia by Evaluating the Change From Baseline in EQ-5D(Euro Quality of Life-5 Dimension) Index Score at Month 12 in the ITT Population.
Description: The Euro Quality of Life - 5 dimension index (EQ-5D) is the result of the application of a formula that essentially attaches values (also called weights) to each of the levels (no, some, or heavy problems) in each dimension (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). These weights are issued from a representative sample of the general population. The total possible maximum value was 1 (healthy life) and the minimum value was 0 (death).
Time Frame: 12 months
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 343 | 360
Scores on a scale | 0.193 (0.0167) | 0.168 (0.0162)

15. Secondary Outcome: To Evaluate the Effect of Quetiapine XR Versus Risperidone at Month 12 in the ITT Population Regarding Health Economics Outcomes by Evaluating the Functional Improvement Rate of the Modified Vocational Status Index/ Location Code Index: Stable State
Description: Stable State was defined as having the same status in occupational and residential status as at Baseline.
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants with stable state
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 268 | 291
Participants with stable state | 160 | 171

16. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone Regarding Health Economics Outcomes by Evaluating the Mean Number of Lost School/Work Days at Month 12 in the ITT Population
Description: Workers and students are defined from the modified vocational status index excluding subjects "Retired" or "Unemployed, whether or not expected to work".
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 158 | 169
Days | 10 (38.54) | 6.7 (30.53)

17. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone Regarding Health Economics Outcomes by Evaluating the Participants With at Least 1 Hospitalization Due to Psychiatric Disorders at Month 12 in the ITT Population
Description: All hospitalizations due to psychiatric disorders during the study (i.e. from Visit 1 to Termination date + 30 days) in inpatients units, in emergency wards, and in day clinics.
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Participants | 37 | 21

18. Secondary Outcome: Number of Subjects Who Had an Unscheduled Visits Due to Worsening of Schizophrenia, Dose Change, or Adverse Event at Month 12 in the ITT Population
Description: Unscheduled visits due to worsening of schizophrenia, dose change or adverse event including the hospitalizations due to psychiatric disorders during the study (i.e. from Visit 1 to Termination date + 30 days) in inpatients units, in emergency wards and in day clinics.
Time Frame: Month 12
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Participants | 94 | 70

19. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone Regarding Health Economics Outcomes by Evaluating the Time Between First Study Drug Intake and First Hospitalization for Patients With 1 Hospitalization in the ITT Population
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 35 | 19
Days | 144.3 (97.14) | 152.8 (87.86)

20. Secondary Outcome: Number of Participants Using Antidepressants at Month 12 in the ITT Population
Description: The number of participants who were taking at least 1 antidepressant at Month 12. Antidepressants are all concomitant medications classified in the Anatomical Therapeutic Chemical(ATC)Subgroup "N06-Antidepressants".
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Participants | 72 | 63

21. Secondary Outcome: The Effect of Quetiapine XR Versus Risperidone Regarding Health Economics Outcomes by Evaluating the Number of Participants Using Other Psychotropic Medications at Month 12 in the ITT Population
Description: Other psychotropic medications include antiepileptics, anti-parkinson drugs, antipsychotics, and antidepressants.
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Participants | 138 | 141

22. Secondary Outcome: The Compliance of Patients Taking Quetiapine XR Versus Risperidone at Month 12 by Evaluating the Number of Participants Who Returned Study Drug at Month 12 in the ITT Population
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 379 | 392
Participants | 270 | 249

23. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Participants With a Treatment-emergent Adverse Event (TEAEs) at Month 12 in the Safety Population
Description: Treatment-emergent adverse events are defined as adverse events that occurred after the first intake of the study medication (or on the same day).
Time Frame: 12 months
Population: The Safety population at Month 12 is presented. For Quetiapine XR, 4 subjects did not take study drug, resulting in 391 evaluable subjects compared with the Randomized population (395 subjects). For Risperidone, 1 subject did not take study drug, results in 402 evaluable subjects compared with the Randomized population (403 subjects).
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 391 | 402
Participants | 238 | 258

24. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Participants Who Discontinued the Study Because of an TEAE at Month 12 in the Safety Population
Description: as for outcome 23
Time Frame: 12 months
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 391 | 402
Participants | 57 | 48

25. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Participants Who Had at Least 1 Extra-pyramidal TEAE at Month 12 in the Safety Population
Description: as for outcome 23
Time Frame: 12 months
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 391 | 402
Participants | 38 | 83

26. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Extra-pyramidal Events at Month 12 in the Safety Population
Description: Extra-pyramidal events include tremor, hypokinesia, muscle rigidity, hyperkinesia, and extrapyramidal disorder.
Time Frame: 12 months
Population: as for outcome 23
Measure: Number; unit: Events
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 391 | 402
Events | 51 | 112

27. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Participants Who Had at Least 1 Cardiac TEAE at Month 12 in the Safety Population
Description: as for outcome 23
Time Frame: 12 months
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 391 | 402
Participants | 22 | 17

28. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Mean Change From Baseline to Month 12 in Prolactin Levels in the Safety Population
Description: The normal range for men is 0 to 14, and for women is 0 to 24.
Time Frame: 12 months
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 332 | 340
ng/mL | -7.735 (32.8559) | 15.990 (46.3367)

29. Secondary Outcome: The Safety and Tolerability of Quetiapine XR vs Risperidone by Evaluating the Number of Participants at Month 12 in Safety Population With Individual Symptoms Assessed by the Modified Udvalg for Kliniske Undersogelser, Side Effect Rating Scale: Neurologic
Description: Symptoms are graded according to degree (not present to severe) and causal relationship (improbable, possible, probable). An individual AE is defined as an AE with a worse degree compared with Baseline and with a possible or probable relationship to study drug.
Time Frame: 12 months
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 209 | 224
Participants | 4 | 20

30. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Participants at Month 12 in the Safety Population With Individual Symptoms Assessed by the Modified UKU: Hyperprolactinaemia in Women
Description: Symptoms are graded according to degree (not present to severe) and causal relationship (improbable, possible, probable). Hyperprolactinaemia in women is defined as number of women who show the individual adverse event (AE) hyperprolactinaemia. An individual AE Hyperprolactinaemia is defined as an AE with a worse degree of hyperprolactinaemia compared with baseline and with a possible or probable relationship to study drug.
Time Frame: Month 12
Population: Safety population at Month 12 is presented. Quetiapine XR: Out of 160 evaluable women, 73 were missing individual AE "Hyperprolactinaemia" data.
  Risperidone: Out of 171 evaluable women, 74 were missing individual AE "Hyperprolactinaemia" data".
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 87 | 97
Participants | 0 | 10

31. Secondary Outcome: The Safety and Tolerability of Quetiapine XR Versus Risperidone by Evaluating the Number of Participants at Month 12 in the Safety Population With Individual Symptoms Assessed by the Modified UKU: Sexual Dysfunction in Men
Description: Symptoms are graded according to degree (not present to severe) and causal relationship (improbable, possible, probable). Sexual dysfunction in men is defined as number of men who show the individual adverse event (AE) sexual dysfunction. An individual AE sexual dysfunction is defined as an AE with a worse degree of sexual dysfunction compared with baseline and with a possible or probable relationship to study drug.
Time Frame: Month 12
Population: Safety population at Month 12 is presented. Quetiapine XR: Out of 231 evaluable men, 111 were missing individual AE "Sexual Dysfunction" data".
  Risperidone: Out of 231 evaluable men, 106 were missing individual AE "Sexual Dysfunction" data".
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Risperidone
Number analyzed (Participants) | 120 | 125
Participants | 9 | 13

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Risperidone
Serious Adverse Events (participants affected / at risk) | 45/391 | 26/402
Other Adverse Events (participants affected / at risk) | 238/391 | 258/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=391) | Risperidone (N=402)
Schizophrenia (Psychiatric disorders) | 12 | 5
Psychotic Disorder (Psychiatric disorders) | 9 | 5
Abnormal Behavior (Psychiatric disorders) | 2 | 1
Acute Psychosis (Psychiatric disorders) | 2 | 1
Agitation (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 1
Suicide Attempt (Psychiatric disorders) | 3 | 0
Aggression (Psychiatric disorders) | 1 | 1
Alcohol Abuse (Psychiatric disorders) | 1 | 1
Schizoaffective Disorder (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
Mental Disorder (Psychiatric disorders) | 1 | 0
Panic Attack (Psychiatric disorders) | 1 | 0
Schizophreniform Disorder (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Brain Stem Stroke (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Extrapyramidal Disorder (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Neuroleptic Malignant Syndrome (Nervous system disorders) | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes Meelitus (Metabolism and nutrition disorders) | 0 | 1
Bone Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary Tumor Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Osteoarthritis (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=391) | Risperidone (N=402)
Somnolence (Nervous system disorders) | 71 | 47
Headache (Nervous system disorders) | 23 | 39
Dizziness Postural (Nervous system disorders) | 23 | 18
Sedation (Nervous system disorders) | 25 | 15
Tremor (Nervous system disorders) | 7 | 29
Insomnia (Psychiatric disorders) | 30 | 52
Anxiety (Psychiatric disorders) | 33 | 38
Tension (Psychiatric disorders) | 18 | 20
Constipation (Gastrointestinal disorders) | 40 | 23
Aptyalism (Gastrointestinal disorders) | 33 | 21
Nausea (Gastrointestinal disorders) | 18 | 26
Asthenia (General disorders) | 22 | 25
Weight Increased (Investigations) | 18 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No